CLINICAL TRIAL: NCT03560973
Title: A Double-blind, Placebo Controlled, Randomized Multicenter Phase II Study Evaluating Gemcitabine With or Without Ramucirumab as II Line Treatment for Advanced Malignant Pleural Mesothelioma
Brief Title: A Double Blind, Placebo Controlled, Randomized Phase II Study Evaluating Gemcitabine With or Without Ramucirumab , for II Line Treatment MPM
Acronym: RAMES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GOIRC-03-2016
Record Dates: First submitted 2018-05-18; First posted 2018-06-19 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2020-07

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Gemcitabine; Ramucirumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gemcitabine + Ramucirumab (Experimental): Gemcitabine 1000 mg/m2 iv D1, D8 plus Ramucirumab 10 mg/kg iv (21 days cycles)
  Interventions: Drug: Gemcitabine; Drug: Ramucirumab
- Gemcitabine + Placebo (Placebo Comparator): Gemcitabine 1000 mg/m2 iv D1, D8 plus placebo (21 days cycles)
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — ramucirumab/ placebo was added to gemcitabine
  Other Names: gemsol
Drug: Ramucirumab — ramucirumab/ placebo was added to gemcitabine
  Other Names: CYRAMZA
  Arms: Gemcitabine + Ramucirumab

SUMMARY:
Study RAMES is a multicentre, double-blind, randomized Phase II study exploring the efficacy and evaluating the safety of the addition of ramucirumab to gemcitabine as the second-line treatment of patients with diffuse pleural mesothelioma. Patients will be randomly assigned (1:1) to receive intravenous gemcitabine 1000 mg/m2 on days 1 and 8 every 21 days with placebo or combined with intravenous ramucirumab 10 mg/Kg (ramucirumab group) on day 1 of a 21 day cycle until PD. Randomisation will be done via a centralized system and will stratified by performance status (0-1 vs 2), age (≤70 vs >70), histology (epithelioid vs others), time to progression (TTP) after a previous treatment (first line therapy, adjuvant or neoadjuvant therapy) (< 6 months vs ≥6 months).

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a histopathologically or cytologically confirmed diagnosis of malignant pleural mesothelioma.
2. The patient has documented disease progression after the last dose of first-line chemotherapy for metastatic disease,

   a. Patients who are intolerant to first-line chemotherapy regimens are eligible. Disease progression must be assessed after the last dose of first-line therapy.
3. The patient received combination chemotherapy prior to disease progression.

   1. Prior chemotherapy regimens must include a platinum or pemetrexed component. Exposure to antineoplastic therapy, in addition to platinum and/or pemetrexed, is acceptable if the agents were used in the first-line metastatic or neoadjuvant/adjuvant setting.
   2. Patients who have had one or more components of first-line chemotherapy discontinued because of toxicity, but continued to receive the other component(s), are eligible following disease progression.
4. The patient has metastatic disease or locally advanced disease that is measurable, or nonmeasurable but evaluable, by radiological imaging per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1) (Eisenhauer et al. 2009 Baseline tumor assessment should be performed using a high resolution computed tomography (CT) scan using intravenous and oral contrast unless clinically contraindicated. Magnetic resonance imaging (MRI) is acceptable if a CT cannot be performed.
5. The patient has an ECOG performance status of 0-2
6. The patient has adequate organ function.
7. The patient is at least 18 years old or of an acceptable age according to local regulations, whichever is older.
8. The patient has provided written informed consent prior to any study-specific procedures and is amenable to compliance with protocol schedules and testing.
9. The patient has an estimated life expectancy of 12 weeks in the judgment of the investigator.
10. The patient has resolution to Grade 1 by Common Terminology Criteria for Adverse Events CTCAE Version 4 NCI 2009, of all clinically significant toxic effects of previous anticancer therapy.
11. The patient, if male, is sterile (including vasectomy confirmed by post-vasectomy semen analysis) or agrees to use a reliable method of birth control and to not donate sperm during the study and for at least 12 weeks following the last dose of study treatment.
12. The patient, if female, is surgically sterile, is postmenopausal, or agrees to use a highly effective method of birth control during the study and for 12 weeks following the last dose of study treatment. A highly effective method of birth control is defined as one that results in a low failure rate when used consistently and correctly.
13. The patient, if female and of child-bearing potential, must have a negative serum or urine pregnancy test within 7 days prior to randomization.

    Exclusion Criteria:
14. The patient has cancer with histology other than mesothelioma.
15. The patient is receiving chronic therapy with any of the following within 7 days prior to randomization:

    1. nonsteroidal anti-inflammatory agents (NSAIDs; such as indomethacin, ibuprofen, naproxen, or similar agents)
    2. other anti-platelet agents (such as clopidogrel, ticlopidine, dipyridamole, or anagrelide) Aspirin use at doses up to 325 mg/day is permitted.
16. The patient received radiotherapy within 14 days prior to randomization. Any lesion requiring palliative radiotherapy or which has been previously irradiated cannot be considered for response assessment.
17. The patient received >1 line of prior therapy for the treatment MPM.
18. The patient received previous treatment with agents targeting the VEGF/VEGF Receptor 2 signaling pathway, including previous exposure to ramucirumab.
19. The patient has documented brain metastases, leptomeningeal disease, or uncontrolled spinal cord compression. Screening of asymptomatic patients is not required.
20. The patient has a significant bleeding disorder or vasculitis or had a Grade 3 bleeding episode within 12 weeks prior to randomization.
21. The patient experienced any arterial thromboembolic event (ATE), including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 6 months prior to randomization.
22. The patient has symptomatic congestive heart failure (CHF; New York Heart Association II-IV) or symptomatic or poorly controlled cardiac arrhythmia.
23. The patient has uncontrolled hypertension, as defined in CTCAE Version 4.0, prior to initiating study treatment, despite antihypertensive intervention. CTCAE Version 4.0 defines uncontrolled hypertension as Grade >2 hypertension; clinically, the patient continues to experience elevated blood pressure (systolic >160 mmHg and/or diastolic >100 mmHg) despite medications).
24. The patient underwent major surgery within 28 days prior to randomization or central venous access device placement within 7 days prior to randomization. The patient has a serious or nonhealing wound, ulcer or bone fracture within 28 days prior to enrollment.
25. The patient has selective or planned major surgery to be performed during the course of clinical trial.
26. The patient has a history of gastrointestinal (GI) perforation or fistula within 6 months prior to randomization.
27. The patient has a history of inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) 12 months prior to randomization.
28. The patient has an acute or subacute bowel obstruction or history of chronic diarrhoea that is considered clinically significant in the opinion of the investigator.
29. The patient has either of the following:

    1. cirrhosis at a level of Child-Pugh B (or worse)
    2. cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites resulting from cirrhosis and requiring ongoing treatment with diuretics and/or paracentesis.
30. The patient has known allergy or hypersensitivity to any components of study treatment.
31. The patient received any previous investigational therapy within 4 half -lives of the investigational agent prior to randomization.
32. The patient has a serious illness or medical condition including, but not limited to, the following:

    1. known human immunodeficiency virus infection or acquired immunodeficiency syndrome-related illness
    2. active or uncontrolled clinically serious infection
33. The patient is pregnant or breast-feeding.
34. The patient has a concurrent active malignancy other than the following:

    1. adequately treated not melanomatous skin cancer
    2. curatively treated in situ carcinoma of the cervix or other not invasive carcinoma or in situ neoplasm A patient with a history of prior malignancy is eligible if he or she has been disease free for 3 years prior to randomization.
35. The patient has a serious nonhealing: (a) wound, (b) peptic ulcer, or (c) bone fracture, within 28 days prior to randomization.
36. The patient experienced any Grade 3 or 4 venous thromboembolic event (VTE) that is considered by the investigator to be life-threatening or that is symptomatic and not adequately treated by anticoagulation therapy, within 6 months prior to randomization (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant")
37. The patient has any condition (for example, psychological, geographical, or medical) that does not permit compliance with the study and follow-up procedures or suggests that the patient is, in the investigator's opinion, not an appropriate candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
OS | 36 months
  time from the date of randomization to the date of death from any cause. gemcitabine with placebo,

SECONDARY OUTCOMES:
PFS | 36 months
  Progression-free survival (PFS) is measured from the date of randomization to the date of radiographic documentation of progression (as defined by RECIST v1.1) or the date of death due to any cause, whichever is earlier. RECIST 1.1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]). | 36 months
  TEAEs, AESIs, SAEs, and hospitalizations, Clinical laboratory tests, vital signs, and physical examinations
ORR | 36 months
  ORR is the proportion of randomized patients achieving a best overall response of complete response (CR) or partial response (PR).
DCR | 36 months
  DCR is the proportion of randomized patients achieving a best overall response of CR, PR, or stable disease (SD).
Predictive molecular markers | 36 months
  polymorphisms associated with ramucirumab response
Quality life | 36 months
  survey completed by patients at cycles
Predictive molecular markers | 36 months
  Evaluation of circulating pro-angiogenic factors in response to Ramucirumab treatment
Predictive molecular markers | 36 months
  Effect of the mutational asset of the tumor on Ramucirumab response

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Pinto, MD, Principal Investigator — Gruppo Oncologico Italiano di Ricerca Clinica
Locations (1):
- Struttura Complessa di OncologiaIRCCS- Istituto in Tecnologie Avanzate e Modelli Assistenziali in Oncologia Arcispedale Santa Maria Nuova, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinto C, Zucali PA, Pagano M, Grosso F, Pasello G, Garassino MC, Tiseo M, Soto Parra H, Grossi F, Cappuzzo F, de Marinis F, Pedrazzoli P, Bonomi M, Gianoncelli L, Perrino M, Santoro A, Zanelli F, Bonelli C, Maconi A, Frega S, Gervasi E, Boni L, Ceresoli GL. Gemcitabine with or without ramucirumab as second-line treatment for malignant pleural mesothelioma (RAMES): a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Oncol. 2021 Oct;22(10):1438-1447. doi: 10.1016/S1470-2045(21)00404-6. Epub 2021 Sep 6. PMID 34499874